CLINICAL TRIAL: NCT05051670
Title: The Safety and Feasibility of Reduced Port Robotic Distal Gastrectomy Using da Vinci SP for Early Gastric Cancer
Brief Title: da Vinci SP Robotic Gastrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2021-0881
Record Dates: First submitted 2021-09-10; First posted 2021-09-21 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Gastric Cancer
Keywords: da vinci SP; robotic surgery; gastrectomy; gastric cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SP group (Experimental): patients group underwent gastrectomy using da vinci SP
  Interventions: Procedure: da vinc SP gastrectomy

INTERVENTIONS:
Procedure: da vinc SP gastrectomy — radical subtotal gastrectomy performed by da vinci SP

SUMMARY:
Laparoscopic surgery revolutionized the surgical treatment of gastric cancer saving large incsion and associated pain. Robotic surgical system was introduced to enhance the minimally invasive surgery using articulating robotic arm. The da vinci SP system, which enables single-port surgery, can allow surgeon to provide radical gastrectomy with minimal scar and associated pain.

DETAILED DESCRIPTION:
This study is a phase 1/2, single-arm surgical clinical trial. The primary endpoint is the safety of da vinci robotic gastrectomy. The secondary endpoint is operative time, bleeding, bowel recovery, and hospital stay. In the clinic, informed consent is received from patient who is scheduled to undergo radical gastrectomy. After the general anesthesia, low midline transverse incision is made at suprapubic area. After inserting SP port into the peritoneal cavity, additional port is inserted via right flank that would be used for assistant's energy device and suction devices. Radical subtotal gastrectomy is perfromed using cardiere-forceps, monopolar scissors, and maryland forceps. Reconstruction after gastrectomy is decided according to surgeon's preference. three days after gastrectomy, if the diet build up is complete and the patients has no evidence of complication, the patient is discharged from the hospital. Four weeks after gastrectomy, the patient will be followed up at the clinic. Major complication event within 30days after gastrectomy will be analyzed as primary endpoint as well as other secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed adenocarcinoma of stomach scheduled to undergo radical gastrectomy
* Between 20-80
* ASA score (American society of anesthesiology) class: I - III
* Signed to informed consent after through explanation about the study

Exclusion Criteria:

* distant metastasis
* EMR/ESD canddiate
* complicated gastric cancer (obstruction or perforation)
* Active other primary tumor
* Vulerable subject (illiterate, pregnant)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-12-11 (Actual)

PRIMARY OUTCOMES:
major complication | 30 days after gastrectomy
  Clavien-Dindo classification grade 3 or more

SECONDARY OUTCOMES:
Operation time | 30 days after gastrectomy
  duation of operation in minutes
bleeding | 30 days after gastrectomy
  amount of bleeding shed during the operation in ml
bowel recovery | 30 days after gastrectomy
  gas passing day after the surgery
Hospital stay | 30 days after gastrectomy
  days between the opeation day to discharge day

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jeong O, Park YK. Clinicopathological features and surgical treatment of gastric cancer in South Korea: the results of 2009 nationwide survey on surgically treated gastric cancer patients. J Gastric Cancer. 2011 Jun;11(2):69-77. doi: 10.5230/jgc.2011.11.2.69. Epub 2011 Jun 30. PMID 22076206
- [Background] Lee JH, Kim KM, Cheong JH, Noh SH. Current management and future strategies of gastric cancer. Yonsei Med J. 2012 Mar;53(2):248-57. doi: 10.3349/ymj.2012.53.2.248. PMID 22318810
- [Background] Kitano S, Iso Y, Moriyama M, Sugimachi K. Laparoscopy-assisted Billroth I gastrectomy. Surg Laparosc Endosc. 1994 Apr;4(2):146-8. PMID 8180768
- [Background] Kim HH, Hyung WJ, Cho GS, Kim MC, Han SU, Kim W, Ryu SW, Lee HJ, Song KY. Morbidity and mortality of laparoscopic gastrectomy versus open gastrectomy for gastric cancer: an interim report--a phase III multicenter, prospective, randomized Trial (KLASS Trial). Ann Surg. 2010 Mar;251(3):417-20. doi: 10.1097/SLA.0b013e3181cc8f6b. PMID 20160637
- [Background] Zeng YK, Yang ZL, Peng JS, Lin HS, Cai L. Laparoscopy-assisted versus open distal gastrectomy for early gastric cancer: evidence from randomized and nonrandomized clinical trials. Ann Surg. 2012 Jul;256(1):39-52. doi: 10.1097/SLA.0b013e3182583e2e. PMID 22664559
- [Background] Kim YM, Baek SE, Lim JS, Hyung WJ. Clinical application of image-enhanced minimally invasive robotic surgery for gastric cancer: a prospective observational study. J Gastrointest Surg. 2013 Feb;17(2):304-12. doi: 10.1007/s11605-012-2094-0. Epub 2012 Dec 1. PMID 23207683
- [Background] Cruz CJ, Huynh F, Kang I, Lee WJ, Kang CM. Initial experiences of robotic SP cholecystectomy: a comparative analysis with robotic Si single-site cholecystectomy. Ann Surg Treat Res. 2021 Jan;100(1):1-7. doi: 10.4174/astr.2021.100.1.1. Epub 2020 Dec 30. PMID 33457391
- [Background] Kang SK, Jang WS, Kim SW, Kim SH, Han SW, Lee YS. Robot-assisted laparoscopic single-port pyeloplasty using the da Vinci SP(R) system: initial experience with a pediatric patient. J Pediatr Urol. 2019 Oct;15(5):576-577. doi: 10.1016/j.jpurol.2019.08.003. Epub 2019 Aug 15. PMID 31570233
- [Background] Gomes MTV, Machado AMN, Podgaec S, Barison GAS. Initial experience with single-port robotic hysterectomy. Einstein (Sao Paulo). 2017 Oct-Dec;15(4):476-480. doi: 10.1590/S1679-45082017AO4134. PMID 29364368
- [Background] Tokunaga M, Sugisawa N, Kondo J, Tanizawa Y, Bando E, Kawamura T, Terashima M. Early phase II study of robot-assisted distal gastrectomy with nodal dissection for clinical stage IA gastric cancer. Gastric Cancer. 2014;17(3):542-7. doi: 10.1007/s10120-013-0293-3. Epub 2013 Sep 5. PMID 24005955
- [Background] Lee S, Kim JK, Kim YN, Jang DS, Kim YM, Son T, Hyung WJ, Kim HI. Safety and feasibility of reduced-port robotic distal gastrectomy for gastric cancer: a phase I/II clinical trial. Surg Endosc. 2017 Oct;31(10):4002-4009. doi: 10.1007/s00464-017-5435-y. Epub 2017 Feb 15. PMID 28205030
- [Background] Park JY, Jo MJ, Nam BH, Kim Y, Eom BW, Yoon HM, Ryu KW, Kim YW, Lee JH. Surgical stress after robot-assisted distal gastrectomy and its economic implications. Br J Surg. 2012 Nov;99(11):1554-61. doi: 10.1002/bjs.8887. PMID 23027072
- [Background] Kim HH, Han SU, Kim MC, Hyung WJ, Kim W, Lee HJ, Ryu SW, Cho GS, Song KY, Ryu SY. Long-term results of laparoscopic gastrectomy for gastric cancer: a large-scale case-control and case-matched Korean multicenter study. J Clin Oncol. 2014 Mar 1;32(7):627-33. doi: 10.1200/JCO.2013.48.8551. Epub 2014 Jan 27. PMID 24470012
- [Background] Tokunaga M, Kondo J, Tanizawa Y, Bando E, Kawamura T, Terashima M. Postoperative intra-abdominal complications assessed by the Clavien-Dindo classification following open and laparoscopy-assisted distal gastrectomy for early gastric cancer. J Gastrointest Surg. 2012 Oct;16(10):1854-9. doi: 10.1007/s11605-012-1981-8. Epub 2012 Jul 31. PMID 22847575
- [Background] Kim SM, Ha MH, Seo JE, Kim JE, Choi MG, Sohn TS, Bae JM, Kim S, Lee JH. Comparison of Reduced Port Totally Laparoscopic Distal Gastrectomy (Duet TLDG) and Conventional Laparoscopic-Assisted Distal Gastrectomy. Ann Surg Oncol. 2015 Aug;22(8):2567-72. doi: 10.1245/s10434-014-4333-y. Epub 2015 Jan 7. PMID 25564174
- [Derived] Park SH, Kim YN, Hwang J, Kim KY, Cho M, Kim YM, Hyung WJ, Kim HI. Safety and feasibility of reduced-port robotic distal gastrectomy for gastric cancer: a phase I/II clinical trial using the da Vinci Single Port(SP) robotic system. Sci Rep. 2023 Oct 30;13(1):18578. doi: 10.1038/s41598-023-45655-6. PMID 37903856